CLINICAL TRIAL: NCT05520034
Title: Effectiveness of Health Education Program Among Patients & Family Caregivers on Modifiable Risk Factors mRS 0 to 4 to Reduce Recurrence of Stroke After Discharge From a Tertiary Hospital in Bangladesh
Brief Title: Reduction of Recurrence of Stroke by Nurse-led Education in Bangladesh
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hiroshima University (Other)
Collaborators: National Institute of Neuro Sciences & Hospital, Bangladesh (Other Government)
Responsible Party: Principal Investigator, Mahabuba Afrin, Doctoral Researcher, Hiroshima University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 151
Record Dates: First submitted 2022-08-23; First posted 2022-08-29 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Stroke
Keywords: Stroke; Caregiver; Recurrence of stroke; Health education; Bangladesh
MeSH Terms: conditions — Stroke; Health Education

STUDY DESIGN:
Intervention Model Description: Randomized control trial (RCT) study
Masking Description: Two-arm open-label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The participants provided health education regarding understanding stroke and the risk factors, lifestyle changes related to modifiable factors, (self)-monitoring of daily blood pressure (BP), and compliance with medication and hospital/clinic visits. At 6 and 12 months RA nurses collected data and samples for lab tests from the patient's house if the patient cannot come to NINSH for any reason. We provided all the patients with lab test costs and transportation fees if they visited any healthcare center for any lab test related to our study.
  Interventions: Behavioral: Health Education
- Control Group (No Intervention): The participants received a one-time telephone call from research nurses every month to keep in contact (telephone calls did not include health education). At 6 and 12 months RA nurses collected data and samples for lab tests from the patient's house if the patient cannot come to NINSH for any reason. We provided all the patients with lab test costs and transportation fees if they visited any healthcare center for any lab test related to our study.

INTERVENTIONS:
Behavioral: Health Education — The participants received a 45mins, face-to-face group health education after enrollment and during the 6th month by a RA nurse. Participants received the same health education over the phone call if the patient and family caregiver could not come for any reason. They also received a digital BP machine, a salt-measurement spoon, a medication box, and a recording notebook for monitoring. The intervention group receives health education above and reminder telephone calls provided by research assistant nurses every month (1st month to 3rd month: twice a month, and 4th month to 12th month: once a month)
  Arms: Intervention group

SUMMARY:
Stroke is a major public issue that can be occurred a patient with severe and unbearable disability for a long time. Recurrence of stroke is increasing due to a lack of knowledge and compliance with treatment regarding the modifiable risk factors of stroke and behavioral and lifestyle changes. Nurse-led health education with (self) monitoring of modifiable risk factors and behaviors can be an effective way to create knowledge about the behavioral changes in stroke patients.

The investigators hypothesized that health education among first stroke patients and their family caregivers could reduce the stroke recurrence rate by controlling modifiable risk factors compared to the first stroke patients without health education.

DETAILED DESCRIPTION:
In Bangladesh, the top cause of death per 100,000 population for both sexes aged all ages in 2019 is stroke. About 79.9 percent of the total patients were suffering from ischemic stroke, and 15.7 percent and 4.6 percent were diagnosed with hemorrhagic and subarachnoid hemorrhage respectively. One study found the cumulative recurrence rate was 14.7% at three months, 15.3% at six months, 17.3% at the ninth month, and 20% at one year (n=150).

This study aims to evaluate the effect of health education among first-stroke patients and their family caregivers for reducing the recurrence of stroke. The investigators also assess the number and rate of all adverse events, changes in values of modifiable risk factors, and change scores in knowledge, lifestyle behavior, medication adherence, and QoL.

In this study, participants were the first stroke patients who were discharged from the National Institute of Neurosciences & Hospital (NINSH) and the family caregivers of the patients. Written informed consent is received from the patient when the patient is the main person of self-management of recurrence prevention, if the patient cannot give consent by disability, his/her family caregiver provided consent.

At baseline, blood specimens such as blood total cholesterol, HDL-cholesterol, HbA1c, and diagnosis including adverse events and blood pressure measurement data were obtained from the hospital records/patient's chart.

At first, the research assistant (RA) nurse should confirm the written consent form for the participants. Then, the RA nurse took the baseline data through the interview. The raw data is stored and locked in secured places in NINSH.

Confidentiality of data is of utmost importance; therefore, every effort is made to safeguard the identity of participants and protect subject privacy. All hard copies of data are stored under lock and kept in the NINSH.

The sample size was based on the calculation of a 10% reduction in recurrence rate compared with the control group with a statistical power of 80% at α= 0.05 (2-tailed). Considering the dropout rate of 10%, the final sample size is 432 (2 arms).

To compare the outcomes of the Intervention Group and Control Group, an intention-to-treat (ITT) analysis and a full analysis set (FAN) were conducted. Descriptive analysis was done to assess the baseline data. For categorical data, the chi-square (X2) test, and for continuous variables, the t-test, or Mann-Whitney U test was employed to compare the two groups where appropriate. For secondary endpoints, after adjusting for confounding variables such as age, an analysis of covariance (ANCOVA) was used to assess the effect of the intervention on the outcomes. To compensate for missing data, the last observation carried forward was measured. The significance level will be set at P=0.05. Data will be analyzed using SPSS (version 26.0; IBM Corp).

In 5% of the study participants, the quality control team independently checked the collected data on the same day using a field-tested methodology. Detected errors were corrected immediately at the field site. The findings of the quality control team are considered for necessary corrections if any major discrepancies are found.

ELIGIBILITY:
For patient

1. Who was discharged from NINSH to home or who visited NINSH right after getting a stroke
2. First-time stroke
3. All types of strokes, except subarachnoid haemorrhage
4. modified Rankin Scale (0 - 4)
5. Stroke patient who is 18 years old and above
6. Both males & females
7. Who provided written consent & willing to participate in the study

For family caregivers

1. Primary caregivers irrespective of sex and aged 18 years old and above, living with the patient who take care of an above patient and who meets all of the inclusion criteria (will be decided by one person)
2. Who will provide written consent & willing to participate in the study

Exclusion Criteria:

Exclusion criteria of patient

1. Who has stroke with the recurrence
2. Stroke subtype: caused by genetic problems or injury/accident
3. Patients with multi-organ failure or terminal stage
4. Participation in other clinical trials
5. Unwillingness to participate in the study
6. Not having a mobile phone at home
7. mRS 5

Exclusion criteria of caregiver

1. Who is not living with the patient
2. Who is under 18 years old
3. Who is mentally unstable and/or cognitively impaired (diagnosed cases)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Estimated)
Dates: Start 2022-10-02 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Change of the recurrence rate of stroke. | 12 months
  Compare the recurrence rate of stroke between the intervention group and the control group

SECONDARY OUTCOMES:
Change of the number of adverse events | 12 months
  Compare the number of all causes of death, and cardiovascular events between the intervention group and the control group. The adverse event refers that all cases that need to be diagnosed: for example, new onset of acute myocardial infarction (AMI) and unstable angina, heart failure (with hospitalization), PAD (peripheral arterial disease: hospitalization)
Change in values of blood pressure level | 12 months
  Compare value of blood pressure (mmHg) between the intervention group and the control group.
Change in value of HbA1c | 12 months
  Compare value of HbA1c (%) between the intervention group and the control group.
Change in non-HDL cholesterol | 12 months
  Compare value of non-HDL cholesterol (mg/dl) (total cholesterol minus HDL cholesterol) between the intervention group and the control group.
Changes in scores in knowledge related to stroke | 12 months
  Compare scores in knowledge related to stroke (the researcher-developed "Knowledge questionnaire of stroke") between the intervention group and the control group. The questionnaire consists of 10 items with "No/Wrong answer", "Yes/Correct answer", and "Don't know" answers. The score ranges from 0-20, and a higher score indicates having better knowledge.
Changes in scores in lifestyle behavior related to stroke | 12 months
  Compare scores in lifestyle behavior related to stroke (the researcher-developed "Lifestyle behavior questionnaire related to stroke") between the intervention group and the control group. The questionnaire consists of 14 items (6 items will not be counted) with a Likert scale with the frequency of behaviors. The score ranges from 0-37, and a higher score indicates having better lifestyle behavior.
Changes in scores in medication adherence | 12 months
  Compare scores of behavior changes in medication adherence measured by a "Medication adherence related questionnaire" between the intervention group and the control group.
  The questionnaire consists of 4 items with "Yes=0" and "No=1" answers. The score ranges from 0-4, and a higher score indicates better compliance.
Changes in scores in QoL | 12 months
  Compare behavior changes in QoL measured by a "WHOQOL- BREF Bangla Version-2 items)" between the intervention group and the control group. Each item scores from 1 (very poor/very dissatisfied) to 5 (very good/very satisfied), and ranges (mean of 2 items) from 1 to 5, a higher mean indicates a better QoL.

CONTACTS AND LOCATIONS:
Overall Officials: KATM Ehsanul Huq, PhD, Principal Investigator — Hiroshima University
Locations (1):
- National Institute of Neurosciences & Hospital, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clarke DJ, Forster A. Improving post-stroke recovery: the role of the multidisciplinary health care team. J Multidiscip Healthc. 2015 Sep 22;8:433-42. doi: 10.2147/JMDH.S68764. eCollection 2015. PMID 26445548
- [Background] Katan M, Luft A. Global Burden of Stroke. Semin Neurol. 2018 Apr;38(2):208-211. doi: 10.1055/s-0038-1649503. Epub 2018 May 23. PMID 29791947
- [Background] GBD 2019 Stroke Collaborators. Global, regional, and national burden of stroke and its risk factors, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet Neurol. 2021 Oct;20(10):795-820. doi: 10.1016/S1474-4422(21)00252-0. Epub 2021 Sep 3. PMID 34487721
- [Derived] Afrin M, Huq KATME, Khan SU, Das SC, Chowdhury MSJH, Fukuoka Y, Fukushima Y, Moriyama M. Effectiveness of a Health Education Program to Reduce Recurrence of Stroke by Controlling Modifiable Risk Factors in a Specialized Hospital in Bangladesh: Randomized Controlled Trial. JMIR Public Health Surveill. 2025 May 27;11:e72233. doi: 10.2196/72233. PMID 40424617
- [Derived] Afrin M, Khan SU, Das SC, Huq KATME, Moriyama M. Effectiveness of a Health Education Program for Patients Who Had a Stroke and Their Caregivers by Controlling Modifiable Risk Factors to Reduce Stroke Recurrence in a Tertiary Hospital in Bangladesh: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Dec 15;12:e51178. doi: 10.2196/51178. PMID 38100172